CLINICAL TRIAL: NCT06094504
Title: Impact of Full Spectrum Light on Outcomes of Infants With Intestinal Failure
Brief Title: Spectral Lighting and Intestinal Failure
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-0566
Record Dates: First submitted 2023-09-21; First posted 2023-10-23 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Intestinal Failure
MeSH Terms: conditions — Intestinal Failure

STUDY DESIGN:
Intervention Model Description: N-of-1 study design in which each subject will serve as their own control.
Masking Description: Data analyst will be blinded as to lighting condition exposure of subject (spectral lighting period vs control lighting period) when analyzed samples were collected.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lighting cycling (Spectral vs Conventional) (Experimental): The study protocol will commence the Monday after study subject enrollment, if medically feasible, and will consist of four weeks of alternating periods of 3 days of daytime conventional (CON) hospital lighting followed by 4 days of daytime full spectrum lighting (FS) including violet and blue light wavelengths.
  Interventions: Other: Spectral Lighting

INTERVENTIONS:
Other: Spectral Lighting — Spectral room lighting containing violet and blue wavelengths of light capable of stimulating non-visual opsins including OPN5 and OPN3.

SUMMARY:
The goal of this exploratory n-of-1-study is to compare markers of metabolism in infants with intestinal failure between two lighting environments. Investigators are seeking to learn whether supplementing the lighting environment of infants with intestinal failure with blue and violet wavelengths of light will allow more efficient utilization of the nutrition provided to participants by influencing hormones involved in regulation of growth and development as compared to a conventional lighting environment.

Pre-clinical studies suggest that violet and blue wavelengths of light are involved in molecular pathways that help regulate metabolic activity.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 32 weeks post-menstrual age (PMA)
* diagnosis or anticipated diagnosis of intestinal failure by qualified provider
* have an anticipated hospital stay of at least 5 weeks following initiation of study participation

Exclusion Criteria:

* Infants with major congenital anomalies outside of the gastrointestinal tract
* Infants with aneuploidy (having an abnormal amount of chromosomes)
* Infants <32 weeks post-menstrual age (PMA)
* Infants who are anticipated to require a major surgery after enrollment other than anastomosis.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
plasma protein concentration of insulin | For four weeks, once a week for each lighting condition and once a week during the predawn hours after each lighting condition, for a total of four samples per week.
  Protein concentrations of plasma insulin as analyzed by SomaScan large scale proteomics assay will be compared among plasma samples taken in lighting conditions and between each lighting condition and dark.
plasma protein concentration of leptin | For four weeks, once a week for each lighting condition and once a week during the predawn hours after each lighting condition, for a total of four samples per week.
  Protein concentrations of plasma insulin as analyzed by SomaScan large scale proteomics assay will be compared among plasma samples taken in lighting conditions and between each lighting condition and dark.

SECONDARY OUTCOMES:
temperature | For the duration of the participant's 4-week study timeline
  body temperature as measured throughout the day, usually every 3-4 hrs
heart rate | For the duration of the participant's 4-week study timeline
  heart rate throughout the day, as collected every 3-4 hrs
Phosphorus concentration | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  concentration of Phosphorus in serum (mg/dL)
Magnesium concentration | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  concentration of Magnesium in serum (mg/dL)
Calcium concentration | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  concentration of Calcium in serum (mg/dL)
Sodium concentration | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  concentration of Sodium in serum (mmol/L)
Potassium concentration | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  concentration of Potassium in serum (mmol/L)
Chloride concentration | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  concentration of Chloride in serum (mmol/L)
glucose | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  glucose concentration in mg/dL
Blood Urea Nitrogen | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  blood urea nitrogen concentration in mg/dL
Creatinine | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  creatinine concentration in mg/dL
Albumin | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  albumin concentration in gm/dL
Total protein level | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  total protein concentration in gm/dL
Alanine Aminotransferase (ALT) | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  Alanine Aminotransferase concentration in unit/L
Aspartate Aminotransferase (AST) | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  Aspartate Aminotransferase (AST) concentration in unit/L
Alkaline Phosphatase (ALP) | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  Alkaline Phosphatase (ALP) concentration in unit/L
Gamma Glutamyl Transferase (GGT) | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  Gamma Glutamyl Transferase (GGT) concentration in unit/L
Triglyceride | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  Triglyceride concentration in mg/dL
Total Bilirubin | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  Total Bilirubin concentration in mg/dL
Direct Bilirubin | Typically collected twice-weekly for the duration of the participant's 4-week study timeline
  Direct Bilirubin concentration in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: James M Greenberg, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Zhang KX, D'Souza S, Upton BA, Kernodle S, Vemaraju S, Nayak G, Gaitonde KD, Holt AL, Linne CD, Smith AN, Petts NT, Batie M, Mukherjee R, Tiwari D, Buhr ED, Van Gelder RN, Gross C, Sweeney A, Sanchez-Gurmaches J, Seeley RJ, Lang RA. Violet-light suppression of thermogenesis by opsin 5 hypothalamic neurons. Nature. 2020 Sep;585(7825):420-425. doi: 10.1038/s41586-020-2683-0. Epub 2020 Sep 2. PMID 32879486
- [Background] Nayak G, Zhang KX, Vemaraju S, Odaka Y, Buhr ED, Holt-Jones A, Kernodle S, Smith AN, Upton BA, D'Souza S, Zhan JJ, Diaz N, Nguyen MT, Mukherjee R, Gordon SA, Wu G, Schmidt R, Mei X, Petts NT, Batie M, Rao S, Hogenesch JB, Nakamura T, Sweeney A, Seeley RJ, Van Gelder RN, Sanchez-Gurmaches J, Lang RA. Adaptive Thermogenesis in Mice Is Enhanced by Opsin 3-Dependent Adipocyte Light Sensing. Cell Rep. 2020 Jan 21;30(3):672-686.e8. doi: 10.1016/j.celrep.2019.12.043. PMID 31968245
- [Background] Tarttelin EE, Bellingham J, Hankins MW, Foster RG, Lucas RJ. Neuropsin (Opn5): a novel opsin identified in mammalian neural tissue. FEBS Lett. 2003 Nov 20;554(3):410-6. doi: 10.1016/s0014-5793(03)01212-2. PMID 14623103
- [Background] Hair AB, Good M. Dilemmas in feeding infants with intestinal failure: a neonatologist's perspective. J Perinatol. 2023 Jan;43(1):114-119. doi: 10.1038/s41372-022-01504-4. Epub 2022 Sep 20. PMID 36127395
- [Background] Gattini D, Roberts AJ, Wales PW, Beath SV, Evans HM, Hind J, Mercer D, Wong T, Yap J, Belza C, Huysentruyt K, Avitzur Y. Trends in Pediatric Intestinal Failure: A Multicenter, Multinational Study. J Pediatr. 2021 Oct;237:16-23.e4. doi: 10.1016/j.jpeds.2021.06.025. Epub 2021 Jun 18. PMID 34153281